CLINICAL TRIAL: NCT05859386
Title: Optimizing Mindfulness-Based Cognitive Therapy Maintenance
Brief Title: Optimizing Mindfulness Based Cognitive Therapy (MBCT) Maintenance
Acronym: OMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Mental Insight Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-37109
Record Dates: First submitted 2023-05-04; First posted 2023-05-16 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Depression
Keywords: depression; mindfulness
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The first group will be a single group aimed at initial intervention refinement. The second group will be randomized to either receive the intervention or enter a wait-list control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness maintenance program (Experimental): Participants receive: (1) Four-week course to strengthen and extend skills learned in 8-week MBCT course, (2) Monthly 1.5 hour meeting session, and (3) Monthly check-in survey.
  Interventions: Behavioral: Mindfulness maintenance program
- Wait-list (No Intervention): Participants receive follow-up measures but no intervention until the end of the wait-list period.

INTERVENTIONS:
Behavioral: Mindfulness maintenance program — 1. Four-week course to strengthen and extend skills learned in 8-week MBCT course. This will consist of four 2-hour sessions, occurring weekly for four weeks.
  2. Monthly 1.5 hour meeting sessions. These will be led by an experienced MBCT teacher and will consist of a group meditation practice, a check-in time, and discussion of a topic relevant to the MBSR course.
  3. Monthly check-in survey. This will be a brief (5 - 10 minute) survey (using Qualtrics) with questions about mood (PROMIS Depression and Positive Affect scales) and recent meditation practice.
  Arms: Mindfulness maintenance program

SUMMARY:
Mindfulness-Based Cognitive Therapy (MBCT) combines meditation practices from Mindfulness-Based Stress Reduction (MBSR) with cognitive behavioral therapy to improve mental health. Although there is evidence that MBCT provides a variety of mental health benefits, it is particularly designed to prevent depression relapse, which occurs in 80% of people with a history of two episodes of depression. MBCT reduces depression relapse rates by 30%, on average after an eight-week course, and has lower relapse rates than continuing antidepressant medication. However, it is unknown what should be done following the program to optimize its long-term benefit. The investigators plan to conduct a pilot study in preparation for larger-scale clinical trial to determine the most effective maintenance approaches once MBCT has ended. The investigators gathered stakeholder input from MBCT graduates and MBCT teachers to inform the development of maintenance programs for MBCT. From this the investigators formulated several components of a maintenance program for MBCT. This includes providing a booster course for people who have already completed the MBCT program. This will be delivered as a 4-week course, meeting weekly, followed by monthly sessions to help participants build self-efficacy and agency with regard to creating their own plan for relapse prevention. This booster course is adapted from a 12-week program developed by Dr. Willem Kuyken at the Oxford Centre for Mindfulness. The team is planning the following sessions: 1 Deepening mindfulness with a focus on interoceptive awareness. 2) Hedonic system: Appreciating the light within. This would focus on positive emotion. 3) Responding not reacting 4) Two themes: taking care of ourselves, taking care of others. Integrating lessons into daily life with regards to sleep, diet, healthy relationships, behavioral activation. The study will also provide monthly follow-up sessions. The current study is a pilot study aimed at refining the intervention, providing initial data on acceptability and feasibility, and preliminary use of outcome measures in the context of the proposed study design.

DETAILED DESCRIPTION:
The current study is a pilot study aimed at refining a maintenance program for MBCT program graduates. It will provide initial data on acceptability and feasibility, and preliminary use of outcome measures in the context of the proposed study design. The first study group aims to have 10 - 15 participants and will be single arm, with the aim of getting feedback to refine the intervention program. The second study group will aim to enroll between 15 and 30 participants, who will be randomized to receive the intervention program or to a wait-list control group (who will receive the 4-week course 4 months later).

Intervention program: The intervention program will have three components that research subjects will be asked to participate in:

Four-week course to strengthen and extend skills learned in 8-week MBCT course. This will consist of four 2-hour sessions, occurring weekly for four weeks. They will cover content that builds on the original 8-week course. These will be led by an experienced teacher trained in leading MBCT courses with a background in mental health. Sessions will be conducted on a video conferencing platform (Zoom). As part of the course, participants will be asked to develop their own depression relapse plan that describes actions they can take that will be helpful if they are becoming depressed.

Monthly 1.5 hour meeting sessions. These will be led by an experienced MBCT teacher and will consist of a group meditation practice, a check-in time, and discussion of a topic relevant to the MBSR course. The monthly sessions will continue for a minimum of 3 months after the end of the last four-week course. Participants from the different four-week courses will join the same monthly meeting sessions. The investigators anticipate that the 2nd four-week course will start about 4 months after the first course, so that participants in the first group will have about 7 monthly meeting sessions.

Monthly check-in survey. This will be a brief (5 - 10 minute) survey (using Qualtrics) with questions about mood (Patient-Reported Outcomes Measurement Information System {PROMIS} Depression and Positive Affect scales) and recent meditation practice. For participants with elevated depression scores, trained study staff will send an email with the participant's earlier depression relapse plan as a reminder, and set a time to check-in with the participant by phone or Zoom to see how they are doing. If indicated, staff can arrange a brief (15 minutes or less) check-in with the monthly session MBCT teacher to go over current steps to prevent depression relapse.

For each of these steps, staff will follow-up with reminders/check-ins if participants unexpectedly miss sessions of the four-week course or monthly meetings, or do not complete the monthly check-in survey. Participants can opt-out at any time if they do not want reminders/check-ins.

Enrollment visit: Participants who may be eligible based on screening survey will be invited to schedule a Zoom visit with study staff to determine final eligibility (primarily rule out high risk fo suicide), learn more about what study participation involves, and review the study consent form. If there are any concerns that arise during this visit, participants will potentially be referred to the Project Director, Dr. Patty Moran, for additional assessment of issues such as suitability for a group intervention.

Baseline and Follow-up Questionnaires: Participants will complete a study questionnaire at baseline (before starting the four-week course), 1 month (end of course), and every 3 months thereafter as long as monthly meetings sessions are occurring for the study ( anticipated to be at 4 months from study start for both groups and 8 months if in the first four-week course). The questionnaire will include standardized measures of decentering, ruminative/repetitive thought, mindfulness, and self-compassion. At follow-up it will include feedback.

Possible Focus Group/Exit Interview: Participants may be invited to participate in an interview or focus group to provide additional feedback about their experience in the program. Interviews and focus groups will take place over Zoom.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. Previously completed MBCT program.
3. A main reason (per self-report) for taking MBCT was for depression

5. Have smartphone or other device for attending virtual classes 6. Ability to speak and read English 7. Lives in US

Exclusion Criteria:

1. Patient Health Questionnaire 8 (PHQ8) score >14 or 5+ items endorsed "more than half the days" or more, one of which corresponds to Question #1 or #2 (generally regarded as indicative of current Major Depressive Disorder).
2. High current risk of suicide on Columbia-Suicide Severity Rating Scale (CSSR-S) or history of attempt in past year
3. Unable or unwilling to attend Zoom group-based sessions as scheduled
4. History of Bipolar 1 disorder, Psychosis or Schizophrenia, or Borderline Personality disorder
5. Substance use, mental health, or other condition that in the opinion of the investigators will make participation in a group setting difficult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Scale (CSQ) scores | 4 months
  Self-assessed satisfaction with care will be measured using the CSQ questionnaire. Scores on the 1979 version of the CSQ questionnaire range from 8 to 32, with higher scores indicating higher levels of satisfaction.

SECONDARY OUTCOMES:
Client Satisfaction Scale (CSQ) scores | 1 month
  Self-assessed satisfaction with care will be measured using the CSQ questionnaire. Scores on the 1979 version of the CSQ questionnaire range from 8 to 32, with higher scores indicating higher levels of satisfaction.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression 8a scores | Baseline to 4 months change
  A change in PROMIS depression 8a scores will be measured during the first four months of the study. The PROMIS depression 8a questionnaire is a self-assessed questionnaire that asks participants to respond to 8 questions with a 5-point ordinal rating scale of "Never," "Rarely," "Sometimes," "Often," and "Always." Questionnaire scores range from 8 to 40, with higher scores indicating a greater severity of depression.
Change in Experiences Questionnaire scores | Baseline to 4 months change
  A change in Experiences Questionnaire scores will be measured during the first four months of the study. The Experiences Questionnaire is a 20-item self-report measure targeting decentering, defined as the ability to observe one's thoughts and feelings as temporary.
  The Experiences Questionnaire is a standardized self-assessed questionnaire that asks participants to respond to 20 questions on a 5-point Likert scale from Never (1) to Always (5). Scores range from 20 to 100, with higher scores indicating greater decentering.
Change in Five Facet Mindfulness Questionnaire-short form (FFMQ-sf) scores | Baseline to 4 months change
  Self-assessed mindfulness will be measured using the Five Facet Mindfulness Questionnaire (FFMQ-15), a 15 question self-report scale that measures mindfulness with regards to thoughts, experiences, and actions in daily life. Items are rated on a 5-point scale of "Never or very rarely true (1)" "Rarely true (2)," "Sometimes true (3)," "Often true (4)," and "Very often or always true (5)."The FFMQ-15 measures 5 facets of mindfulness: Observing, Describing, Acting with Awareness, Non-judgement, and Non-reactivity. Total scores range from 15-60. Subscale or facet scores range from 3-15. Higher scores reflect greater mindfulness.
Change in Self-Compassion Scale-Short Form (SCS-sf) scores | Baseline to 4 months change
  Self-compassion will be measured with the Self-compassion Scale-Short Form (SCS-SF), a 12-item measure of how often one behaves kindly and caringly towards oneself in difficult life situations. Participants respond on a five-point Likert scale (1 = 'Almost never' to 5 = 'Almost always'). Total scale scores range from 12 to 60, with higher scores reflective of greater self-compassion.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Hecht, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No